CLINICAL TRIAL: NCT04333888
Title: BrainBoost - A Neurofeedback Booster for Emotion Regulation Therapy
Brief Title: A Neurofeedback Booster for Emotion Regulation Therapy
Acronym: BrainBoost
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Paret (Other)
Collaborators: Yale University (Other); AE Foundation (Other)
Responsible Party: Sponsor-Investigator, Christian Paret, Principal Investigator, Central Institute of Mental Health, Mannheim
Organization: Central Institute of Mental Health, Mannheim (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-513N
Record Dates: First submitted 2020-03-26; First posted 2020-04-03 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Neurofeedback

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Behavioral: Neurofeedback
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Neurofeedback — fMRI neurofeedback training of amygdala downregulation
  Arms: Treatment

SUMMARY:
This is a proof-of-concept study that aims to test the additional value of adjuvant neurofeedback treatment for psychotherapy. Three sessions of real-time fMRI neurofeedback will be administered to N=22 patients with BPD while they receive residential Dialectical Behavior Therapy treatment. In addition, outcomes are assessed from a control group with same sample size who do not receive the treatment.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 BPD diagnosis
* informed consent
* EtOH and tox negative on the day of neurofeedback
* BSL-23 score >=1.87 at DBT halftime

Exclusion Criteria:

* pharmacotherapy with opiates
* standing benzodiazepines (bedtime-only benzodiazepines and anti-histamines allowed)
* pregnancy
* epilepsy
* life-time diagnosis schizophrenia or bipolar disorder I
* significant current or past neurological illness
* BMI<16.5
* usual safety criteria for magnetic resonance imaging

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in affective instability | Before treatment, immediately after treatment + follow-up measure (3 months)
  Mean successive squared differences (MSSD) of six-item negative affect scale measured via behavioural sampling using ecological momentary assessment (EMA) over four days. MSSD will be compared between baseline and post-treatment timepoints.

SECONDARY OUTCOMES:
Change in emotion regulation | Before treatment, immediately after treatment + follow-up measure (3 months)
  Negative and neutral pictures are either presented with instruction to regulate or to respond naturally (view). BOLD response in the amygdala (and the rest of the brain) is measured and subjective ratings of regulation success are collected. Changes (between the time points) in differences of the two conditions (regulate vs. view) are measured for both: amygdala BOLD response and subjective ratings of regulation success.
Change in borderline symptomatology | Before treatment, immediately after treatment + 2 follow-up measures (3 months, 6 months)
  Facets of BPD are assessed with questionnaires, including impulsivity. Borderline Symptom List (BSL-23) score will be used for assesment of BPD symptoms. This scale has 23 items, each scored 0-4, and total score is mean item endorsement (sum of all items divided by 23). Higher scores indicate more symptom endorsement.
Change in resting state brain connectivity | Before treatment, immediately after treatment + follow-up measure (3 months)
  Patients get a 10 min brain scan (fMRI) without active task. Data are analysed to compare changes in intrinsic functional brain connectivity (BOLD activation of amygdala with other brain regions) during resting state before and after neurofeedback training.
Change in amygdala reactivity | Before treatment, immediately after treatment + follow-up measure (3 months)
  Patients will perform a task, in which blocks of faces with negative emotional expressions and scrambled pictures will be presented. This task leads to considerable amygdala activation. With this task, we want to observe effects of neurofeedback on spontaneous amygdala activation.
Structural changes in the brain | Before the first neurofeedback training and after the last neurofeedback training
  By including DTI sequences before and after the neurofeedback intervention, we want to explore changes in FA/fiber structure of the brain. (exploratory analysis)

CONTACTS AND LOCATIONS:
Locations (1):
- Central Institute of Mental Health, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zaehringer J, Ende G, Santangelo P, Kleindienst N, Ruf M, Bertsch K, Bohus M, Schmahl C, Paret C. Improved emotion regulation after neurofeedback: A single-arm trial in patients with borderline personality disorder. Neuroimage Clin. 2019;24:102032. doi: 10.1016/j.nicl.2019.102032. Epub 2019 Oct 16. PMID 31795041